CLINICAL TRIAL: NCT01708083
Title: Polymorphids and mRNA Expression in Genes, Significant for Developing Obesity and Typ II Diabetes in Different Types/Localisations of Fat Tissue
Brief Title: Polymorphids an mRNA Expression in Obese Genes
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Associated professor, MD, Karolinska Institutet
Other Study IDs: 2009/1629-31/3
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Polymorphism; mRNA Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsys; Fat from oment, thigh and abdomen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Type 2 Diabetes and BMI>35: Patients with type 2 diabetes and body mass index 35 or more.
- BMI>35: Patients undergoing surgery, gastric bypass or cholecystectomy, without diabetes type 2 and body mass index 35 or more
- BMI 18-27: Patients undergoing surgery, cholecystectomy or reflux, without type 2 diabetes and body mass index between 18-27

SUMMARY:
Fat tissue from omenta, thigh and abdomen taken under anesthesia on subjects undergoing laparoscopic surgery, cholecystectomy, reflux surgery or gastric by-pass (GBP).

Are there any difference in polymorphids and/or mRNA expression in genes significant for developing obesity, between normal weight and obese individuals, with or without diabetes typ 2 .

Are there any difference in polymorphids and/or mRNA expression in different types of fat tissue

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* laparoscopic surgery (Gastric by-pass, cholecystectomy, antireflux surgery)
* Normal weight without type 2 diabetes BMI 18-25
* Obese without type 2 diabetes BMI>35
* Obese with type 2 diabetes BMI>35

Exclusion Criteria:

* under 18 years
* open surgery
* pregnancy
* BMI >27-<35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tree groups; group I: diabetes type II with BMI>35 Group II: no diabetes BMI>35 Group III: no diabetes BMI 18-27
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Differences in polymorphids and/or mRNA expression in genes, significant for developing obesity and type 2 diabetes, between patients with normal weight and obesity | approximatly 30 minutes after start of operation
  fat biopsy taken from abdomen, omenta and thigh at surgery
Difference in polymorphids and/or mRNA expression in different types of fat tissue in patients with normal weight or obesity with or without diabetes type 2 | approximatly 30 minutes after start of operation
  fat biopsy; abdomen, omenta and thigh taken at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Ass. prof., Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Ersta hospital, Stockholm, Stockholm County Council
  - Karolinska Institutet, CMM, Stockholm